CLINICAL TRIAL: NCT03383263
Title: Prospective Multi-Center Observational Study to Assess Persistence, Adherence and Changes in Disease Activity in the Children Population of Juvenile Arthritis Patients Treated With Adalimumab (HUMIRA) in the Routine Clinical Settings in the Russian Federation (PETITE)
Brief Title: A Study to Assess Persistence, Adherence and Changes in Disease Activity in the Children Population of Juvenile Arthritis Patients Treated With Adalimumab (HUMIRA®)
Acronym: PETITE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P17-164
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Polyarticular Juvenile Arthritis
Keywords: Humira®; polyarticular juvenile arthritis; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with juvenile arthritis: Children with diagnosed polyarticular juvenile arthritis according to International League of Associations for Rheumatology (ILAR) criteria treated with HUMIRA (adalimumab) in the routine clinical settings in the Russian Federation

SUMMARY:
The objective of this study is to assess persistence, adherence and changes in disease activity in the children population of juvenile arthritis patients treated with adalimumab (HUMIRA®) in the routine clinical settings in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of polyarticular Juvenile Idiopathic Arthritis (JIA) according to International League of Associations for Rheumatology (ILAR) criteria .
* Planned treatment with HUMIRA according to the local product label and prescription guidelines. Alternatively, subjects assigned to HUMIRA treatment not more than 1 month prior to inclusion can be enrolled.
* Negative result of tuberculosis (TB) screening procedure and TB specialist permission to start biologic therapy.
* Patient's informed consent form signed by the parent or guardian/and by the child, if applicable.

Exclusion Criteria:

* Has contraindications for the treatment with HUMIRA according to the latest version of the locally approved label.
* Any biologic drugs taken prior to 3 months of enrolment in the study.
* Patients treated with any biosimilar version of HUMIRA
* Previous participation and dropout from this study.
* Patients participating in another clinical and/or observational study priory 3 months before the enrolment to this study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with diagnosed polyarticular juvenile arthritis according to ILAR criteria treated with HUMIRA (adalimumab) in routine clinical settings in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Assessing Humira persistence | Up to 30 days after the last dose of the study drug (approximately 52 weeks)
  Persistence is defined as the time (in days) between the start date of HUMIRA (adalimumab) treatment and the earliest date of discontinuation of Humira (adalimumab) or drop out of study, or lost to follow up.

SECONDARY OUTCOMES:
Proportion of patients with Humira adherence | Up to Week 48 of treatment
  The adherence to Humira will be assessed.
Proportion of patients with 30% American College of Rheumatology (ACR) pediatric responses | Up to Week 48 of treatment
  It is defined as 30% improvement respectively in a minimum of three core set criteria with worsening of one variable by no more than 30%.
Proportion of patients with 50% American College of Rheumatology (ACR) pediatric responses | Up to Week 48 of treatment
  It is defined as 50% improvement respectively in a minimum of three core set criteria with worsening of one variable by no more than 30%.
Proportion of patients with 70% American College of Rheumatology (ACR) pediatric responses | Up to Week 48 of treatment
  It is defined as 70% improvement respectively in a minimum of three core set criteria with worsening of one variable by no more than 30%.
Change from baseline in physician overall disease activity | From Week 0 to Week 48 of the treatment period
  This is measured using Visual Analog Scale (VAS).
Change from baseline in patient (if appropriate in age) or parent overall well-being | From Week 0 to Week 48 of the treatment period
  This is measured using Visual Analog Scale (VAS).
Assessing Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI) score | Up to 48 weeks of the treatment period
  Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI) score is assessed.
Change from baseline in number of joints with active arthritis | From Week 0 to Week 48 of the treatment period
  The change in number of joints with active arthritis is assessed.
Change from baseline in number of joints with limited range of motion | From Week 0 to Week 48 of the treatment period
  The change in number of joints with limited range of motion is assessed.
Change from baseline in Erythrocyte Sedimentation Rate (ESR) | From Week 0 to Week 48 of the treatment period
  The Erythrocyte Sedimentation Rate is assessed.
Change from baseline in 10-joint Juvenile Arthritis Disease Activity Score (JADAS10) | From Week 0 to Week 48 of the treatment period
  10-joint Juvenile Arthritis Disease Activity Score is assessed.
Proportion of patient with low diseases activity (1.1 - 2 score) | Up to 48 weeks of the treatment period
  This is assessed based on JADAS10 score.
Proportion of patient with moderate disease activity (2.1 - 4.2 score) | Up to 48 weeks of the treatment period
  This is assessed based on JADAS10 score.
Proportion of patients with missed dosed of HUMIRA | Up to 48 weeks of the treatment period
  The proportion of patients with missed dosed of HUMIRA is assessed.
Proportion of patients with predefined Extra-articular manifestations (EAMs) | Up to 48 weeks of the treatment period
  The proportion of patients with predefined EAMs is assessed.
Proportion of patients with any comorbidity | Up to 48 weeks of the treatment period
  Patients with any comorbidities are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (14):
- Russia (14):
  - Republican Children's Clinical Hospital /ID# 204830, Ufa, Bashkortostan Republic
  - Chelyabinsk Regional Children's Clinical Hospital /ID# 204829, Chelyabinsk, Chelyabinsk Oblast
  - Saratov State Medical University n.a. V.I. Razumovskiy /ID# 206319, Saratov, Saratov Oblast
  - Kazan State Medical Academy /ID# 207004, Kazan'
  - Morozovskaya Children's City Clinical Hospital /ID# 207006, Moscow
  - Sechenov First Moscow Medical /ID# 207005, Moscow
  - State Budgetary Healthcare Institution Moscow Region "Moscow Regional Consultati /ID# 212874, Mytischi
  - GBUZ NO Regional Children's Clinical Hospital /ID# 212362, Nizhny Novgorod
  - Privolzhsky Federal Medical Research Center /ID# 206318, Nizhny Novgorod
  - Regional Children's Clinical Hospital /ID# 206121, Orenburg
  - Saint Petersburg State Pediatric Medical University /ID# 203169, Saint Petersburg
  - Samara Regional Clinical Cardiology Clinic /ID# 206120, Samara
  - Federal State Budgetary Educational Institution of Higher Education National Re /ID# 212361, Saransk
  - State Budgetary Health Institution "Regional Children's Clinical Hospital №1" /ID# 212363, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/adalimumab_P17-164.pdf